CLINICAL TRIAL: NCT02216071
Title: A Phase 3, Randomized, Double-Blind, Active-Controlled, Parallel-Group Study of the Comparative Efficacy and Safety of EXL CDOS in Subjects With Acute Otitis Externa
Brief Title: Comparative Efficacy and Safety of Ciprofloxacin 0.3% and Dexamethasone 0.1% in Acute Otitis Externa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exela Pharma Sciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EXL CDOS-300 AOE
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2020-09

CONDITIONS: Acute Otitis Externa
MeSH Terms: interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciprodex®, RLD (Active Comparator): Ciprodex®, Otic Suspension, Twice daily for 7 days
  Interventions: Drug: Ciprodex®
- EXL CDOS (Experimental): EXL CDOS (Ciprofloxacin 0.3% and Dexamethasone 0.1%) Sterile Otic Suspension, Otic Suspension, Twice daily for 7 days
  Interventions: Drug: EXL CDOS (Ciprofloxacin 0.3% and Dexamethasone 0.1%) Sterile Otic Suspension

INTERVENTIONS:
Drug: Ciprodex® — Treatment of acute otitis externa (AOE) when administered twice daily for 7 days
  Arms: Ciprodex®, RLD
Drug: EXL CDOS (Ciprofloxacin 0.3% and Dexamethasone 0.1%) Sterile Otic Suspension — Treatment of acute otitis externa (AOE) when administered twice daily for 7 days
  Other Names: Ciprofloxacin 0.3% and Dexamethasone 0.1% Sterile Otic Suspension
  Arms: EXL CDOS

SUMMARY:
The purpose of the study is to demonstrate the clinical therapeutic non-inferiority of EXL CDOS to commercially available Ciprofloxacin 0.3% and Dexamethasone 0.1% Sterile Otic Suspension (Ciprodex®, Alcon) in the treatment of acute otitis externa (AOE) when administered twice daily for 7 days.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, active-controlled, parallel-group study in adults and children (age 6 months and older) with a diagnosis of AOE with a 2-day screening period followed by a 2-week participation period. Subjects were administered study drug, EXL CDOS or RLD, 4 drops in the affected ear(s) BID for 7 days. The primary endpoint, the proportion of subjects with a clinical AOE score of 0, was measured at the TOC Visit on Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 6 months of age and over;
2. Clinically documented AOE consistent with the diagnostic guidelines of the American Academy of Otolaryngology-Head and Neck Surgery Foundation in 1 or both ears;
3. Inflammation and/or edema ≥2 on the AOE scale, and otorrhea and/or tenderness present;
4. AOE of <4 weeks duration;
5. Intact tympanic membrane(s) in the treated ear(s);
6. Willingness to refrain from swimming through the TOC/ Visit 5;
7. For subjects with AOE associated with hearing aid use, willingness to discontinue the use of hearing aid(s) in the affected ear(s) through the TOC/Visit 5;
8. Ability to complete the study in compliance with the protocol;
9. For adult subjects, ability to understand and provide written informed consent; and
10. For pediatric subjects, a parent or legal guardian has provided written informed consent; and
11. For children age 6 and above, ability to understand and provide assent according to institutional requirements.

Exclusion Criteria:

1. Acute or chronic suppurative otitis media;
2. Post-tympanostomy tube acute otorrhea;
3. Malignant otitis externa;
4. Suspected or overt fungal or viral ear infection;
5. Congenital abnormalities or obstructive bony exostoses of the external auditory canal of the treated ear(s);
6. Seborrheic dermatitis or other dermatologic conditions of the external auditory canal of the treated ear(s) which could confound evaluation;
7. Mastoiditis or other suppurative infectious or non-infectious disorders of the treated ear(s);
8. Malignant tumors of the external auditory canal of the treated ear(s);
9. History of otologic surgery of the treated ear(s), with the exception of tympanic membrane surgery >6 months prior to Baseline;
10. Four or more episodes of otitis externa (OE) in the previous year;
11. Uncontrolled diabetes mellitus;
12. Immunosuppressive disorder, including known Human Immunodeficiency Virus infection;
13. Renal insufficiency;
14. Hepatitis or hepatic insufficiency;
15. Receipt of systemic antibiotic concurrently or within 72 hours prior to Baseline;
16. Receipt of topical otic antibiotic within 24 hours prior to Baseline;
17. Use of systemic corticosteroid concurrently or within 30 days prior to Baseline;
18. Use of topical otic corticosteroids concurrently or within 7 days prior to Baseline;
19. Concurrent use of systemic or topical otic nonsteroidal or other anti-inflammatory drugs;
20. Use of topical vinegar, alcohol, or other astringent otic preparations concurrently or within 24 hours prior to Baseline;
21. Pregnancy, planned pregnancy, or lactation;
22. Known sensitivity or intolerance to quinolone antibacterial agents;
23. Previous participation in this trial;
24. Participation in another investigational drug or vaccine trial concurrently or within 30 days; or
25. Significant acute or chronic medical, neurologic, or psychiatric illness in the subject or parent/guardian that, in the judgment of the Principal Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2014-07-20 (Actual); Primary Completion 2015-08-11 (Actual); Study Completion 2015-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Chair — BioStrategics Consulting Ltd
Locations (48):
- United States (46):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Desert Clinical Research/Clinical Research Advantage, Inc., Mesa, Arizona
  - Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Southland Clinical Research Center, Anaheim, California
  - Southland Clinical Reseach Center, Bellflower, California
  - Alessi Institute, Beverly Hills, California
  - American Clinical Trials, Buena Park, California
  - MCS Clinical Trials, Los Angeles, California
  - Sacramento Ear, Nose and Throat Surgical and Medical Group, Inc, Sacramento, California
  - Benchmark Research, Sacramento, California
  - Clinix Health Services of Colorado/Clinical Research Advantage, Inc., Centennial, Colorado
  - Colorado ENT & Allergy, Colorado Springs, Colorado
  - Colorado Springs Health Partners/Clinical Research Advantage, Inc., Colorado Springs, Colorado
  - Direct Helpers Medical Center, Hialeah, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Abel & Buchheim PR, Inc., Miami, Florida
  - Integrity Clinical Trials, LLC, Miami, Florida
  - Pediatrics & Adolescent Medicine, PA, Marietta, Georgia
  - Urban Family Practice/Clinical Research Advantage, Marietta, Georgia
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Horizon Research Group, LLC, Eunice, Louisiana
  - Woburn Pediatric Associates, Woburn, Massachusetts
  - Pioneer Clinical Research, Bellevue, Nebraska
  - Clinical Research Center for Nevada, LLC, Las Vegas, Nevada
  - ProMetrix Clinical Studies, Morganville, New Jersey
  - Whitehouse Station Family Medicine, Whitehouse Station, New Jersey
  - Asheboro Research Associates, Asheboro, North Carolina
  - Piedmont Ear, Nose, and Throat Associates, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Research Across America, Dallas, Texas
  - Gulf Coast Medical Research, Houston, Texas
  - Gulf Coast Medical Research, Missouri City, Texas
  - Benchmark Research, San Angelo, Texas
  - Mercury Clinical Research, Inc, Splendora, Texas
  - Gulf Coast Medical Research, Sugar Land, Texas
  - Ericksen Research & Development, Clinton, Utah
  - J. Lewis Research/First Med East, Salt Lake City, Utah
  - J. Lewis Research/Foothill Family Clinic South, Salt Lake City, Utah
  - Chyrsalis Clinical Research, St. George, Utah
  - Pi-Coor Clinical Research, LLC, Burke, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Heugenot Pediatrics, PC, Midlothian, Virginia
  - Zain Research, LLC, Richland, Washington
- Puerto Rico (2):
  - Advance Medical Concepts, PSC, Cidra
  - Clinical Research Puerto Rico, San Juan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciprodex®, RLD | EXL CDOS
Started | 254 | 245
Completed | 239 | 233
Not Completed | 15 | 12
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 3 | 5
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprodex®, RLD | EXL CDOS | Total
Number analyzed (Participants) | 254 | 245 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (24.50) | 33.1 (23.54) | 33.2 (24.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 131 | 263
  Male | 122 | 114 | 236
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 81 | 85 | 166
  Not Hispanic or Latino | 173 | 160 | 333
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 16 | 26 | 42
  White | 233 | 210 | 443
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 18 | 15 | 33
  United States | 236 | 230 | 466

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure of AOE
Description: The primary efficacy endpoint was the clinical cure of AOE, defined as the proportion of subjects with a clinical AOE score of 0 at the TOC Visit. Subjects with AOE in both ears were considered to have achieved clinical cure of AOE if the clinical AOE score was 0 for both ears. The clinical AOE score was defined as the sum of scores for inflammation and edema (0=absent, 1=mild, 2=moderate, 3=severe) and tenderness and otorrhea (0=absent, 1=present).
Time Frame: 7 days after the completion of therapy; at Day 15 (+/- 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprodex®, RLD | EXL CDOS
Number analyzed (Participants) | 254 | 245
Participants | 190 | 191

2. Secondary Outcome: Number of Participants With Microbiological Cure (MC)
Description: The secondary efficacy endpoint was the microbiological cure of AOE, defined as the proportion of subjects with microbiological cure at the TOC Visit. Subjects with AOE in both ears were considered to have achieved microbiological cure if microbiological cure was achieved in both ears.
Time Frame: 7 days after the completion of therapy; at Day 15 (+/- 1 day)
Population: The number of participants analyzed represents Bacteria-Positive cohort of subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprodex®, RLD | EXL CDOS
Number analyzed (Participants) | 160 | 149
Participants | 115 | 117

3. Other Pre Specified Outcome: Number of Participants With Adverse Events
Description: Safety outcomes evaluated
  * AEs
Time Frame: Each monitoring visit through 15 +/- 1 days
Population: 499 subjects were randomized as the ITT population, 245 in the EXL CDOS arm & 254 in the RLD arm. All were included in the safety population, but randomization was modified for 36 subjects in the EXL CDOS arm and 43 subjects in the RLD arm to account for available supply of study drug, making 252 subjects in the EXL CDOS arm & 247 in the RLD arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprodex®, RLD | EXL CDOS
Number analyzed (Participants) | 247 | 252
Participants | 60 | 67

ADVERSE EVENTS:
Description: 499 subjects were randomized as the ITT population, 245 in the EXL CDOS arm & 254 in the RLD arm. All were included in the safety population, but randomization was modified for 36 subjects in the EXL CDOS arm and 43 subjects in the RLD arm to account for available supply of study drug, making 252 subjects in the EXL CDOS arm & 247 in the RLD arm.
Arm/Group | Ciprodex®, RLD | EXL CDOS
Serious Adverse Events (participants affected / at risk) | 0/247 | 1/252
Other Adverse Events (participants affected / at risk) | 47/247 | 42/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprodex®, RLD (N=247) | EXL CDOS (N=252)
TMJ Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 — A 41-year-old woman with a history of lupus, was hospitalized with lupus-associated Tempero Mandibular Joint TMJ syndrome with a lupus flare-up at 2 days after beginning study drug treatment. The SAE, which was deemed to be unrelated to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprodex®, RLD (N=247) | EXL CDOS (N=252)
Ear and labyrinth disorder (Ear and labyrinth disorders) | 18 | 15 — Ear discomfort, Ear pruritus, Otorrhoea, Ear Congestion, Ear haemorrhage, Ear swelling, Eustachian tube dysfunction, Excessive cerumen production, Hearing impaired, Tympanic membrane disorder, Tympanic membrane hyperaemia, Ear pain, External ear diso
Photophobia (Eye disorders) | 0 | 1
Gastrointestinal (Gastrointestinal disorders) | 1 | 2
General disorder and administration site conditions (General disorders) | 3 | 1 — Pyrexia, Facial pain, Pain
Infections and Infestations (Infections and infestations) | 13 | 18 — Otitis externa, Otitis media, Sinusitis, Gastroenteritis viral, Candida infection, Conjuctivitis, Herpes zoster, Localised infection, Nasopharyngitis, Pharyngitis, Sepsis, Upper respiratory tract infection, Ear infection fungal, Fungal infection
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 | 3 — Arthropod bite, Hand fracture, Overdose, Concussion, Contusion Laceration, Lip Injurey, Skin abrasion
Heart rate increased (Investigations) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 | 2 — Arthralgia, Temporomandibular joint syndrome, Back pain, Musculoskeletal pain
Nercous system disorders (Nervous system disorders) | 5 | 5 — Headache, Dizziness, Hypoaesthesia, Presyncope, Sinus headache
Respiratory, thoracid and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 3 — Cough, Dyspnoea, Epistaxis, Oropharyngeal pain, Rhinitis allergic, Rhinorrhoea
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 4 — Rash, Dermatitis contact
Menarche (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes